CLINICAL TRIAL: NCT00918892
Title: Assessment of Candidate Protein Expression in Human Breast Cancer Specimens
Brief Title: Assessment of Candidate Protein Expression in Breast Cancer Specimens
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE1108
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer; triple-negative breast cancer; HER2-negative breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gene Expression Profiling; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Previously collected breast cancer tissue samples (paraffin embedded blocks) and normal adjacent tissue are used for immunohistochemistry studies of expression of candidate genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: gene expression analysis — Previously collected breast cancer tissue samples (paraffin embedded blocks) and normal adjacent tissue are used for immunohistochemistry studies of expression of candidate genes.
Other: immunohistochemistry staining method — Previously collected breast cancer tissue samples (paraffin embedded blocks) and normal adjacent tissue are used for immunohistochemistry studies of expression of candidate genes.
Other: laboratory biomarker analysis — Previously collected breast cancer tissue samples (paraffin embedded blocks) and normal adjacent tissue are used for immunohistochemistry studies of expression of candidate genes.

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor tissue samples from patients who have undergone surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if candidate genes display differential expression between normal and cancer breast tissues.

OUTLINE: Previously collected breast cancer tissue samples (paraffin embedded blocks) and normal adjacent tissue are used for immunohistochemistry studies of expression of candidate genes.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Tissue samples available
* Samples are selected based on presence or absence of tumor receptors, (i.e.; estrogen, progesterone, and HER2 receptors) and grouped into following 4 categories:

  * Estrogen receptor (ER)-positive/progesterone receptor (PR)-positive/HER2-negative
  * ER-positive/PR-positive/ HER2-positive by FISH
  * ER-negative/PR-negative/HER2-positive
  * ER-negative/PR-negative/HER2-negative(triple negative or basal-type cancers)

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Exclusion Criteria:

* There are no exclusion criteria in this protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously collected breast cancer tissue samples (paraffin embedded blocks) and normal adjacent tissue are used for immunohistochemistry studies of expression of candidate genes.
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Differential expression of candidate genes between normal and cancer breast tissues | non-applicable
  Approximately 5 slides of each tumor will be collected to provide sufficient samples for replicate staining, if necessary, as well as a staining for a positive control

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Avril, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case1108